CLINICAL TRIAL: NCT06140680
Title: The Effectiveness of the LifelongU Intervention in Habit, Automatic Affective Evaluations and Physical Activity Among University Students With Physical Inactivity
Brief Title: Intervention in Habit, Automatic Affective Evaluations and Physical Activity Among University Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Dandan Huang, Phd Candidate, Universiti Sains Malaysia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DANDAN HUANG
Record Dates: First submitted 2023-11-09; First posted 2023-11-20 (Actual); Last update posted 2023-11-20 (Actual); Status verified 2023-11

CONDITIONS: Physical Inactivity; Sedentary Behavior
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LifelongU (Experimental): Four modules that performed face-to-face physical education lessons:
  1. health-related fitness knowledge
  2. fitness test and training
  3. motor skill training
  4. behavior change techniques (habit formation and implementation intention)
  Interventions: Behavioral: LifelongU
- Physical education (Active Comparator): Classic physical education lessons: physical fitness training and skill training
  Interventions: Behavioral: Physical education

INTERVENTIONS:
Behavioral: LifelongU — The LifelongU intervention is an abbreviation name from LifelongU: Cultivating Physical Literacy for University & Beyond. "LifelongU" is a unique and coined term that symbolizes the program's commitment to promoting physical literacy as a lifelong journey. It combines the words "Lifelong" and "University" to represent an intervention that focuses on physical literacy development not only during the university years but also throughout a person's entire life. The name is designed to convey the idea that physical literacy is an asset that will benefit individuals in all aspects of life, even after they leave the university.
  Arms: LifelongU
Behavioral: Physical education — The control group received 12-week traditional physical education lesson as usual.
  Arms: Physical education

SUMMARY:
The goal of this clinical trial is to test the effectiveness of the LifelongU intervention in habit, automatic affective evaluation and physical activity among university students. The main questions aim to answer are:

* What is the difference in habit, automatic affective evaluation and physical activity between the intervention and control groups?
* What is the difference in habit, automatic affective evaluation and physical activity between the before and after intervention?

Participants will attend 12 sessions of four modules that performed face-to-face physical education lessons. Lesson content included 10-min health-related fitness knowledge, 30-min fitness test and training, 50-min motor skill training with behavior change techniques (90 min per a lesson, once a week).

Researchers will compare control group to see if any effect difference.

DETAILED DESCRIPTION:
A range of behavior change techniques derived from habit formation and self-regulation domain strategies will be used. These include behavioral rehearsal/practice, prompts/cues, and self-monitoring. The overall aim was to help students increase perceptions of physical competence and confidence, build positive affective attitude of physical activity, and develop autonomous association between physical activity and cues of time or events. Moreover, this intervention used student-centered learning strategies, game-centered approach in terms of mode of learning, and flexible in choice of timing, frequency, duration, and intensity of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-25 years
* failure meeting the recommended physical activity guidelines (< 150 minutes MVPA or < 70 minutes VIPA in total a week) at the time of recruitment, screened via the Global Physical Activity Questionnaire

Exclusion Criteria:

* student athletes
* the presence of health conditions that prevented safe engagement in physical activity, screened via the PAR-Q+.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-02-12 (Estimated); Primary Completion 2024-05-17 (Estimated); Study Completion 2024-06-14 (Estimated)

PRIMARY OUTCOMES:
Physical Activity | Assessments will be conducted at baseline (after the screening), 6th week after the baseline, 12th week, and 16th week.
  Using [Global Physical Activity Questionnaire]: the minimum time are 0 minutes per a day and maximum time are 1440 minutes per a day, and higher scores mean a better physical activity level.
Habit | Assessments will be conducted at baseline (after the screening), 6th week after the baseline, 12th week, and 16th week.
  Using questionnaire [Physical activity self-report habit index]: This is a 12-item questionnaire answered on a 7-point Likert scale ranging from 1 (Strongly disagree) to 7 (Strongly agree), with higher scores indicating stronger habit strength.
Association Affective Evaluation | Assessments will be conducted at baseline (after the screening), 6th week after the baseline, 12th week, and 16th week.
  Using [Single-Category Implicit Association Test]: the minimum value is 0 and maximum values is 5, and higher scores mean a positive affective attitude.

CONTACTS AND LOCATIONS:
Locations (1):
- Dandan Huang, Chongqing, Chongqing Municipality, China